CLINICAL TRIAL: NCT03904134
Title: Clinical Transplant-Related Long-term Outcomes of Alternative Donor Allogeneic Transplantation (BMT CTN 1702)
Acronym: BMT CTN 1702
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 1702; 5U24HL138660-02 (NIH); N00014-18-1-2888 (Other Grant/Funding Number: Office of Naval Research)
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Non-hodgkin Lymphoma; Hodgkin Lymphoma; Acquired Aplastic Anemia; Sickle Cell Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: The primary comparison for the interventional study will be between two arms based on biologic assignment, analyzed on an intention-to-treat basis: Arm 1: Patients who are Very Likely to find a matched unrelated donor (MUD), defined as having a >90% chance of finding an 8/8 HLA-matched unrelated donor, for whom a fully matched unrelated donor will be pursued; and Arm 2: Patients who are Very Unlikely to find a MUD, defined as having a <10% chance of finding an 8/8 HLA-matched unrelated donor, for whom a haploidentical, cord blood, or mismatched unrelated donor transplant will be pursued. Patients with a Less Likely chance of finding a MUD, i.e., those not falling into the other two groups (a 26% chance), will be enrolled onto the observational component of the study and analyzed for all relevant endpoints but will not be included in the primary comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Donor Search Prognosis: MUD Very Likely (Other): Patients who are Very Likely to find a matched unrelated donor (MUD), defined as having a >90% chance of finding an 8/8 HLA-matched unrelated donor, for whom a fully matched unrelated donor will be pursued.
  Interventions: Other: Donor Search Prognosis Score
- Donor Search Prognosis: MUD Very Unlikely (Other): Patients who are Very Unlikely to find a MUD, defined as having a <10% chance of finding an 8/8 HLA-matched unrelated donor, for whom a haploidentical, cord blood, or mismatched unrelated donor transplant will be pursued.
  Interventions: Other: Donor Search Prognosis Score
- Donor Search Prognosis: MUD Less Likely (Other): Patients with a Less Likely chance of finding a MUD, i.e., those not falling into the other two groups (a 26% chance), will be enrolled onto the observational component of the study and analyzed for all relevant endpoints but will not be included in the primary comparison.
  Interventions: Other: Donor Search Prognosis Score

INTERVENTIONS:
Other: Donor Search Prognosis Score — Patients will be placed on a study arm after receiving a Donor Search Prognosis Score, which is based on HLA allele frequencies and race/ethnicity. This score predicts the likelihood of successfully identifying a 10/10 matched unrelated donor.Worse search prognosis is associated with racial and ethnic minority status but not with other patient and disease biology characteristics that might influence the success of hematopoietic cell transplantation (HCT). Thus, the use of donor search prognosis in this trial as a tool for biologic assignment to matched unrelated donors vs. mismatched donors provides a mechanism to minimize bias from disease characteristics.

SUMMARY:
The purpose of this study is to determine if a search strategy of searching for an HLA-matched unrelated donor for allogeneic transplantation if possible then an alternative donor if an HLA-matched unrelated donor is not available versus proceeding directly to an alternative donor transplant will result in better survival for allogeneic transplant recipients within 2 years after study enrollment.

DETAILED DESCRIPTION:
This is a multicenter, interventional and observational study to understand factors affecting the likelihood of transplantation in patients without a human leukocyte antigen (HLA) matched family donor and to compare outcomes associated with pursuing an HLA-identical unrelated versus other alternative donor graft sources. Alternative donors are defined as any donor other than an HLA-matched or 1 antigen-mismatched related donor. Patients with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), myelodysplastic syndromes (MDS), Non-Hodgkin lymphoma (NHL), Hodgkin lymphoma (HL), acquired aplastic anemia (AA) or sickle cell disease (SCD) are eligible. The primary comparison for the interventional study will be between two arms based on biologic assignment, analyzed on an intention-to-treat basis: Arm 1: Patients who are Very Likely to find a matched unrelated donor (MUD), defined as having a >90% chance of finding an 8/8 HLA-matched unrelated donor, for whom a fully matched unrelated donor will be pursued; and Arm 2: Patients who are Very Unlikely to find a MUD, defined as having a <10% chance of finding an 8/8 HLA-matched unrelated donor, for whom a haploidentical, cord blood, or mismatched unrelated donor transplant will be pursued. Patients with a Less Likely chance of finding a MUD, i.e., those not falling into the other two groups (a 26% chance), will be enrolled onto the observational component of the study and analyzed for all relevant endpoints but will not be included in the primary comparison.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling the inclusion criteria will be eligible for enrollment in this study. Of those who consent, only patients who lack a suitable HLA-identical or 1 allele or antigen mismatched related donors are evaluable. Patients with an HLA-identical sibling or 1 allele or antigen mismatched family member donor are evaluable as long as the center deems the family member donor as unsuitable for other reasons. Patients may co-enroll with other interventional or observational studies.

1. Patients of all ages with AML, ALL, MDS, NHL, HL, AA, or SCD are eligible.
2. Any planned conditioning regimen and GVHD prophylaxis approach is eligible.
3. Patients must be considered suitable allogeneic transplant candidates at the time of enrollment based on medical history, physical examination, and available laboratory tests. Specific testing for organ function is not required for eligibility but, if available, these tests should be used by the treating physician to judge transplant suitability.
4. Patient and physician must intend to proceed with allogeneic HCT within the next 6 months if a suitable donor is identified.
5. Center plans to follow the algorithm for alternative donor identification: (a) for subjects who are Very Likely to find a MUD, attempt to identify a matched unrelated donor; (b) for a subjects who are Very Unlikely to find a MUD, proceed expeditiously to a haploidentical, cord blood or mismatched unrelated donor.
6. Signed informed consent, and assent if applicable. Consent may be signed prior to completion of family typing but patients will only be considered evaluable upon confirmation that there is no suitable HLA-identical or 1 allele or antigen mismatched related donor available.

Exclusion Criteria:

1. Prior allogeneic HCT (prior autologous transplant is allowed)
2. Previous formal unrelated donor search

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1753 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival for MUD Very Likely and MUD Very Unlikely Arms | 2 years
  Compare overall survival between Very Likely to find a matched unrelated donor search prognosis patients and Very Unlikely to find a matched unrelated donor search prognosis patients who are evaluable.

SECONDARY OUTCOMES:
Cumulative Incidence of Transplant by Donor Search Prognosis Score | 2 years
  To estimate and compare the cumulative incidence of receiving a transplant according to donor search prognosis, regardless of donor search prognosis
Barriers to Transplant | 2 years
  To describe barriers to achieving transplantation with different donor search strategies, regardless of donor search prognosis

OTHER OUTCOMES:
Overall survival in patients transplanted for malignant diseases | 2 years
  To compare overall survival in patients transplanted for malignant diseases, according to the donor search prognosis and the alternative donor used.
Relapse in patients transplanted for malignant diseases | 2 years
  To compare relapse in patients transplanted for malignant diseases, according to the donor search prognosis and the alternative donor used.
Disease-free survival in patients transplanted for malignant diseases | 2 years
  To compare disease-free survival, treatment-related mortality, and acute and chronic GVHD in patients transplanted for malignant diseases, according to the donor search prognosis and the alternative donor used.
Treatment-related mortality in patients transplanted for malignant diseases | 2 years
  To compare treatment-related mortality in patients transplanted for malignant diseases, according to the donor search prognosis and the alternative donor used.
Acute and chronic GVHD in patients transplanted for malignant diseases | 2 years
  To compare acute and chronic GVHD in patients transplanted for malignant diseases, according to the donor search prognosis and the alternative donor used.
Survival in patients with acquired aplastic anemia and sickle cell disease after transplantation | 2 years
  To describe survival in patients with acquired aplastic anemia and sickle cell disease after transplantation, according to the donor search prognosis and the alternative donor used.
Acute and chronic GVHD in patients with acquired aplastic anemia and sickle cell disease after transplantation | 2 years
  To describe acute and chronic GVHD in patients with acquired aplastic anemia and sickle cell disease after transplantation, according to the donor search prognosis and the alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - QoL | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to compare QOL, according to the donor search prognosis and alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - primary graft failure | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of primary graft failure, according to the donor search prognosis and alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - chronic GVHD | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of chronic GVHD, according to the donor search prognosis and alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - time until off systemic immunosuppression | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe time until off systemic immunosuppression, according to the donor search prognosis and alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - GRFS | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of acute grade III-IV and chronic GVHD requiring immunosuppression-free, relapse-free survival (GRFS), according to the donor search prognosis and alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - CRFS | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of moderate-severe chronic GVHD relapse-free survival (CRFS), according to the donor search prognosis and alternative donor used.
AML or ALL in first complete remission or early stage MDS Substudy - current CRFS | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of current CRFS (still on systemic treatment for cGVHD), according to the donor search prognosis and alternative donor used.
QOL Substudy - number of hospital days | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the number of hospital days in the first 100 post-transplant days, according to the donor search prognosis and alternative donor used.
QOL Substudy - infections | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of infections, according to the donor search prognosis and alternative donor used.
QOL Substudy - immune reconstitution | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the incidence of immune reconstitution, according to the donor search prognosis and alternative donor used.
QOL Substudy - late effects after transplantation | 2 years
  In patients with AML or ALL in first complete remission or early stage MDS treated with a limited subset of conditioning and GVHD prophylaxis regimens and transplanted with either matched unrelated donors or haploidentical related donors (QOL Substudy), to describe the late effects after transplantation, according to the donor search prognosis and alternative donor used.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Lee, MD, MPH, Study Chair — Fred Hutchinson Cancer Center; Stefan Ciurea, MD, Study Chair — M.D. Anderson Cancer Center
Locations (52):
- United States (52):
  - City of Hope, Duarte, California
  - University of California, San Diego Medical Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center - Adults, Omaha, Nebraska
  - University of Nebraska Medical Center - Pediatrics, Omaha, Nebraska
  - Rosewell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03904134/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03904134/ICF_001.pdf